CLINICAL TRIAL: NCT02224703
Title: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy and Safety of Cannabidiol (GWP42003-P) in Children and Young Adults With Dravet Syndrome.
Brief Title: GWPCARE2 A Study to Investigate the Efficacy and Safety of Cannabidiol (GWP42003-P) in Children and Young Adults With Dravet Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWEP1424; 2014-002939-34 (EudraCT Number)
Record Dates: First submitted 2014-08-21; First posted 2014-08-25 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Epilepsy; Dravet Syndrome
Keywords: Cannabidiol; CBD; GWP42003-P; Epidiolex
MeSH Terms: conditions — Epilepsy; Epilepsies, Myoclonic | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 10 mg/kg/day GWP42003-P (Experimental): GWP42003-P oral solution (100 mg/milliliter [mL] cannabidiol in sesame oil with anhydrous ethanol with added sweetener [sucralose] and strawberry flavoring). The 10 mg/kg/day dose was defined as 50% of the 20 mg/kg/day dose.
  Interventions: Drug: GWP42003-P
- 20 mg/kg/day GWP42003-P (Experimental): GWP42003-P oral solution (100 mg/mL cannabidiol in sesame oil with anhydrous ethanol with added sweetener [sucralose] and strawberry flavoring). The 20 mg/kg/day dose was recommended by the DSMC after assessment of safety and pharmacokinetic data from Part A of study GWEP1332 (NCT02091206).
  Interventions: Drug: GWP42003-P
- Placebo Control (Placebo Comparator): Excipients only. Participants were pooled from 2 placebo cohorts, half receiving 10 mg/kg/day dose-volume equivalent and half receiving 20 mg/kg/day dose-volume equivalent.
  Interventions: Drug: Placebo Control

INTERVENTIONS:
Drug: GWP42003-P
  Other Names: Cannabidiol; CBD; Epidiolex
  Arms: 10 mg/kg/day GWP42003-P; 20 mg/kg/day GWP42003-P
Drug: Placebo Control
  Other Names: Placebo
  Arms: Placebo Control

SUMMARY:
To investigate the potential antiepileptic effects of cannabidiol (GWP42003-P) in children and young adults with Dravet syndrome.

DETAILED DESCRIPTION:
This study was a 2:2:1:1 randomized, double-blind, 14-week comparison of two dose levels of GWP42003-P (10 milligram/kilogram [mg/kg]/day and 20 mg/kg/day) versus placebo (10 mg/kg/day dose-volume equivalent and 20 mg/kg/day dose-volume equivalent; presented as pooled placebo in the study). A 28-day screening period prior to randomization (to establish baseline parameters) preceded the treatment period, which consisted of a 2-week titration period followed by a 12-week maintenance period. The study aimed to determine the efficacy, safety, and tolerability of GWP42003-P compared with placebo. 20 mg/kg/day was recommended by the Data Safety Monitoring Committee (DSMC) after assessment of safety and pharmacokinetic data from Part A of study GWEP1332 (NCT02091206). The first participant did not enroll into this study until the DSMC reviewed the safety data from Part A of study GWEP1332 (NCT02091206).

Following study completion, all participants were invited to continue to receive GWP42003-P in a separate open-label extension study (GWEP1415; NCT02224573).

ELIGIBILITY:
Key Inclusion Criteria:

* Participant must have been male or female, aged between 2 and 18 years (inclusive).
* Participant must have had a documented history of Dravet syndrome that was not completely controlled by current antiepileptic drugs.
* Participant must have been taking 1 or more antiepileptic drugs at a dose that had been stable for at least 4 weeks.
* All medications or interventions for epilepsy (including ketogenic diet and vagus nerve stimulation) must have been stable for 4 weeks prior to screening and participant was willing to maintain a stable regimen throughout the study.

Key Exclusion Criteria:

* Participant had clinically significant unstable medical conditions other than epilepsy.
* Participant had clinically relevant symptoms or a clinically significant illness in the 4 weeks prior to screening or randomization, other than epilepsy.
* Participant was currently using or had in the past used recreational cannabis, medicinal cannabis, or synthetic cannabinoid-based medications (including Sativex®) within the 3 months prior to study entry and was unwilling to abstain for the duration for the study.
* Participant had any known or suspected hypersensitivity to cannabinoids or any of the excipients of the investigational medicinal products.
* There were plans for the participant to travel outside their country of residence during the study.
* Any history of suicidal behavior or any suicidal ideation of type four or five on the Columbia-Suicide Severity Rating Scale (Children's) at screening.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 199 (Actual)
Dates: Start 2015-04-13 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (23):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Los Angeles, California
  - Sacramento, California
  - Hartford, Connecticut
  - Miami, Florida
  - Savannah, Georgia
  - Chicago, Illinois
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Saint Paul, Minnesota
  - St Louis, Missouri
  - Omaha, Nebraska
  - Lebanon, New Hampshire
  - Buffalo, New York
  - Chapel Hill, North Carolina
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Austin, Texas
  - Fort Worth, Texas
  - Richmond, Virginia
  - Seattle, Washington
- Australia (2):
  - Heidelberg
  - Randwick
- Ramat Gan, Israel
- Netherlands (2):
  - Heeze
  - Zwolle
- Poland (3):
  - Krakow
  - Lodz
  - Warsaw
- Spain (5):
  - Barcelona
  - Madrid
  - Pamplona
  - Seville
  - Valencia

REFERENCES:
- [Derived] Madan Cohen J, Checketts D, Dunayevich E, Gunning B, Hyslop A, Madhavan D, Villanueva V, Zolnowska M, Zuberi SM. Time to onset of cannabidiol treatment effects in Dravet syndrome: Analysis from two randomized controlled trials. Epilepsia. 2021 Sep;62(9):2218-2227. doi: 10.1111/epi.16974. Epub 2021 Jul 15. PMID 34265088
- [Derived] Miller I, Scheffer IE, Gunning B, Sanchez-Carpintero R, Gil-Nagel A, Perry MS, Saneto RP, Checketts D, Dunayevich E, Knappertz V; GWPCARE2 Study Group. Dose-Ranging Effect of Adjunctive Oral Cannabidiol vs Placebo on Convulsive Seizure Frequency in Dravet Syndrome: A Randomized Clinical Trial. JAMA Neurol. 2020 May 1;77(5):613-621. doi: 10.1001/jamaneurol.2020.0073. PMID 32119035

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 43 sites screened participants and 38 sites (23 in the United States, 7 in Spain, 3 in Poland, 2 in Australia, 1 in Israel, and 2 in the Netherlands) randomized participants into the trial. Two sites selected (1 in Israel and 1 in the United States) did not screen any participants.
Pre-assignment Details: To assess eligibility, participants, 2-18 years of age with Dravet syndrome had to be taking 1 or more antiepileptic drugs at a dose which had been stable; and medicated for epilepsy for at least 4 weeks were screened. A total of 285 participants were screened, of which 199 were randomized.
Groups:
- 10 mg/kg/Day GWP42003-P: GWP42003-P oral solution (100 milligrams/milliliter [mg/mL] cannabidiol in sesame oil with anhydrous ethanol with added sweetener [sucralose] and strawberry flavoring). The 10 mg/kilogram (kg)/day dose was defined as 50% of the 20 mg/kg/day dose.
- 20 mg/kg/Day GWP42003-P: GWP42003-P oral solution (100 mg/mL cannabidiol in sesame oil with anhydrous ethanol with added sweetener [sucralose] and strawberry flavoring).The 20 mg/kg/day dose was recommended by the Data Safety Monitoring Committee (DSMC) after assessment of safety and pharmacokinetic data from Part A of study GWEP1332 (NCT02091206).
Period: Overall Study
Arm/Group | 10 mg/kg/Day GWP42003-P | 20 mg/kg/Day GWP42003-P | Placebo Control
Started | 67 | 67 | 65
Received at Least 1 Dose of Study Drug | 66 | 67 | 65
Safety Analysis Set (Received at least 1 dose of study drug and analyzed as per actual treatment received) | 64 (Two participants assigned to the 10 mg/kg/day dose were included in the 20 mg/kg/day group) | 69 (Two participants assigned to the 10 mg/kg/day dose were included in the 20 mg/kg/day group) | 65
Intent to Treat (ITT) Analysis Set (Randomized, received study drug, and had post-baseline efficacy data) | 66 | 67 | 65
Completed | 64 | 61 | 65
Not Completed | 3 | 6 | 0
Not completed — Adverse Event | 0 | 5 | 0
Not completed — Withdrawn by investigator | 1 | 0 | 0
Not completed — Advised by medical monitor | 1 | 0 | 0
Not completed — Withdrawn by parent/guardian | 0 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 10 mg/kg/Day GWP42003-P: GWP42003-P oral solution (100 mg/mL cannabidiol in sesame oil with anhydrous ethanol with added sweetener [sucralose] and strawberry flavoring). The 10 mg/kg/day dose was defined as 50% of the 10 mg/kg/day dose.
- Total: Total of all reporting groups
Arm/Group | 10 mg/kg/Day GWP42003-P | 20 mg/kg/Day GWP42003-P | Placebo Control | Total
Number analyzed (Participants) | 64 | 69 | 65 | 198
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.169 (4.1744) | 9.245 (4.3792) | 9.617 (4.5757) | 9.343 (4.3626)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 32 | 34 | 104
  Male | 26 | 37 | 31 | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 4 | 5
  Black or African American | 1 | 0 | 4 | 5
  White | 55 | 66 | 55 | 176
  Other | 8 | 2 | 1 | 11
Region of Enrollment [Number; unit: participants]
  Australia | 6 | 4 | 3 | 13
  Israel | 0 | 1 | 2 | 3
  Netherlands | 9 | 7 | 9 | 25
  Poland | 8 | 11 | 6 | 25
  Spain | 12 | 14 | 13 | 39
  United States | 29 | 32 | 32 | 93

OUTCOME MEASURES:

1. Primary Outcome: Change In Convulsive Seizures During The Treatment Period Compared To Baseline
Description: Convulsive seizures were defined as tonic-clonic, tonic, clonic, or atonic. Participants or their caregivers recorded the number and type of convulsive seizures each day from screening until completion of dosing using an interactive voice response system (IVRS) diary. The primary endpoint was analyzed using negative binomial regression on the sum of the convulsive seizure counts during the treatment period, based on the ITT analysis set. Baseline included all available data prior to Day 1. Data reported as the ratio of geometric least squares mean in convulsive seizures and expressed as a percentage reduction.
Time Frame: Baseline to Day 99 or Early Termination (ET)
Population: Intention-to-treat (ITT) analysis set: All participants who were randomized and dosed in the trial and had post-baseline efficacy data.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: percentage reduction
Groups:
- 10 mg/kg/Day GWP42003-P: GWP42003-P oral solution (100 mg/mL cannabidiol in sesame oil with anhydrous ethanol with added sweetener [sucralose] and strawberry flavoring). The 10 mg/kg/day dose was defined as 50% of the 20 mg/kg/day dose.
Arm/Group | 10 mg/kg/Day GWP42003-P | 20 mg/kg/Day GWP42003-P | Placebo Control
Number analyzed (Participants) | 66 | 67 | 65
percentage reduction | 48.7 [37.9 to 57.6] | 45.7 [34.2 to 55.2] | 26.9 [11.9 to 39.4]
Statistical Analysis 1: Comparison: 20 mg/kg/Day GWP42003-P vs Placebo Control; Model includes total number of seizures as a response variable and age group, time (baseline and treatment period), treatment, and treatment by time interaction as fixed effects, and participant as a random effect. Log-transformed number of days in which seizures were reported by period is included as an offset. Null hypothesis was that the ratio of GWP42003-P to placebo would be 1; Test type: Superiority; p = 0.0299, Negative binomial regression; Treatment Ratio = 0.743, 95% CI 2-sided [0.568 to 0.971]
Statistical Analysis 2: Comparison: 10 mg/kg/Day GWP42003-P vs Placebo Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0095, Negative binomial regression; Treatment Ratio = 0.702, 95% CI 2-sided [0.538 to 0.916]

2. Secondary Outcome: Change In Total Seizures During The Treatment Period Compared To Baseline
Description: Total seizures were defined as the combination of convulsive and non-convulsive seizures. Convulsive seizures were defined as tonic-clonic, tonic, clonic, or atonic seizures. Non-convulsive seizures were defined as myoclonic, countable partial, other partial, or absence seizures. Participants or their caregivers recorded the number and type of convulsive seizures and non-convulsive seizures each day from screening until completion of dosing using an IVRS diary. Change compared to baseline was calculated as per the primary outcome measure. Data reported as the ratio of geometric least squares mean in total seizures and expressed as a percentage reduction.
Time Frame: Baseline to Day 99 or ET
Population: as for outcome 1
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: percentage reduction
Arm/Group | 10 mg/kg/Day GWP42003-P | 20 mg/kg/Day GWP42003-P | Placebo Control
Number analyzed (Participants) | 66 | 67 | 65
percentage reduction | 56.4 [47.8 to 63.6] | 47.3 [36.9 to 56.0] | 29.7 [16.0 to 41.1]
Statistical Analysis 1: Comparison: 20 mg/kg/Day GWP42003-P vs Placebo Control; Model includes total number of seizures as a response variable and age group, time (baseline and treatment period), treatment, and treatment by time interaction as fixed effects, and participant as a random effect. Log-transformed number of days in which seizures were reported by period is included as an offset; Test type: Superiority; p = 0.0255, Negative binomial regression; Treatment Ratio = 0.749, 95% CI 2-sided [0.581 to 0.965]
Statistical Analysis 2: Comparison: 10 mg/kg/Day GWP42003-P vs Placebo Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0003, Negative binomial regression; Treatment Ratio = 0.620, 95% CI 2-sided [0.481 to 0.799]

3. Secondary Outcome: Participants With A ≥50% Reduction From Baseline In Convulsive Seizure Frequency During The Treatment Period
Description: Convulsive seizures were defined as tonic-clonic, tonic, clonic, or atonic. Participants or their caregivers recorded the number and type of convulsive seizures each day from screening until completion of dosing using an IVRS diary. Baseline included all available data prior to Day 1 (28-day average). Percentage change from baseline was calculated as: ([frequency during the treatment period - frequency during baseline]/frequency during baseline) x 100. The frequency during each period was based on 28-day averages and calculated as: (number of seizures in the period/number of reported days in the IVRS period) x 28. Baseline included all available data prior to Day 1 (28-day average).
Time Frame: Baseline to Day 99 or ET
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg/kg/Day GWP42003-P | 20 mg/kg/Day GWP42003-P | Placebo Control
Number analyzed (Participants) | 66 | 67 | 65
Participants | 29 | 33 | 17
Statistical Analysis 1: Comparison: 20 mg/kg/Day GWP42003-P vs Placebo Control; Test type: Superiority; p = 0.0069, Cochran-Mantel-Haenszel; P-value calculated from a Cochran-Mantel-Haenszel test stratified by age group (2-5, 6-12, and 13-18 years); Odds Ratio (OR) = 2.74, 95% CI 2-sided [1.32 to 5.70]
Statistical Analysis 2: Comparison: 10 mg/kg/Day GWP42003-P vs Placebo Control; Test type: Superiority; p = 0.0332, Cochran-Mantel-Haenszel; P-value calculated from a Cochran-Mantel-Haenszel test stratified by age group (2-5, 6-12, and 13-18 years); Odds Ratio (OR) = 2.21, 95% CI 2-sided [1.06 to 4.62]

4. Secondary Outcome: Caregiver Global Impression Of Change (CGIC) At The Last Visit
Description: On Day 1 (prior to receiving study drug), the caregiver was asked to write a brief description of the participant's overall condition as a memory aid for the CGIC questionnaire at subsequent visits. The CGIC questionnaire comprised the following question, to be rated on a 7-point scale: Since your child started treatment, please assess the status of your child's overall condition (comparing their condition now to their condition before treatment) using the scale below. The markers were: "Very Much Improved"; "Much Improved"; "Slightly Improved"; "No Change"; "Slightly Worse"; "Much Worse"; "Very Much Worse". The CGIC response/score, recorded at each visit, was summarized, on both a categorical and continuous scale, by treatment group. The scores at the last scheduled visit (not including the end of taper or safety follow-up visits) at which participant's last evaluation was performed were analyzed using ordinal logistic regression.
Time Frame: Baseline to Last Visit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 10 mg/kg/Day GWP42003-P | 20 mg/kg/Day GWP42003-P | Placebo Control
Number analyzed (Participants) | 66 | 66 | 65
Participants
  Very Much Improved | 13 | 11 | 1
  Much Improved | 11 | 10 | 8
  Slightly Improved | 21 | 19 | 18
  No Change | 18 | 17 | 32
  Slightly Worse | 2 | 5 | 4
  Much Worse | 1 | 3 | 2
  Very Much Worse | 0 | 1 | 0
Statistical Analysis 1: Comparison: 20 mg/kg/Day GWP42003-P vs Placebo Control; Test type: Superiority; p = 0.0279, Regression, Logistic; Odds Ratio (OR) = 2.02, 95% CI 2-sided [1.08 to 3.78] — Proportional odds modelling was carried out by including treatment group as a fixed factor. The estimated OR tested the null hypothesis that OR was equal to 1
Statistical Analysis 2: Comparison: 10 mg/kg/Day GWP42003-P vs Placebo Control; Test type: Superiority; p = 0.0009, Regression, Logistic; Odds Ratio (OR) = 2.93, 95% CI 2-sided [1.56 to 5.53] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: From Day 1 to Day 137.
Description: Safety Analysis Set: Received at least 1 dose of study drug and were analyzed per treatment received. Two participants randomized to receive GWP42003-P 10 mg/kg/day titrated above the target dose and were therefore assigned to the GWP42003-P 20 mg/kg/day group for all safety analyses.
Arm/Group | 10 mg/kg/Day GWP42003-P | 20 mg/kg/Day GWP42003-P | Placebo Control
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/69 | 0/65
Serious Adverse Events (participants affected / at risk) | 13/64 | 17/69 | 10/65
Other Adverse Events (participants affected / at risk) | 56/64 | 60/69 | 58/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg/kg/Day GWP42003-P (N=64) | 20 mg/kg/Day GWP42003-P (N=69) | Placebo Control (N=65)
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 0
Drug interaction (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0
Status epilepticus (Nervous system disorders) | 5 | 7 | 8
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 3 | 0 | 1
Somnolence (Nervous system disorders) | 2 | 0 | 0
Seizure cluster (Nervous system disorders) | 1 | 0 | 2
Unresponsive to stimuli (Nervous system disorders) | 1 | 0 | 0
Psychogenic seizure (Psychiatric disorders) | 1 | 0 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pneumonia (Infections and infestations) | 3 | 2 | 0
Viral infection (Infections and infestations) | 1 | 1 | 0
Coxsackie viral infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Adenovirus infection (Infections and infestations) | 1 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 10 mg/kg/Day GWP42003-P (N=64) | 20 mg/kg/Day GWP42003-P (N=69) | Placebo Control (N=65)
Diarrhoea (Gastrointestinal disorders) | 11 | 18 | 8
Vomiting (Gastrointestinal disorders) | 4 | 11 | 4
Pyrexia (General disorders) | 15 | 14 | 11
Fatigue (General disorders) | 5 | 14 | 7
Nasopharyngitis (Infections and infestations) | 4 | 8 | 5
Upper respiratory tract infection (Infections and infestations) | 3 | 4 | 3
Urinary tract infection (Infections and infestations) | 0 | 4 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 4 | 0
Alanine aminotransferase increased (Investigations) | 3 | 8 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 8 | 0
Gamma-glutamyltransferase increased (Investigations) | 4 | 4 | 3
Decreased appetite (Metabolism and nutrition disorders) | 10 | 19 | 11
Somnolence (Nervous system disorders) | 14 | 16 | 9
Convulsion (Nervous system disorders) | 3 | 4 | 4
Tremor (Nervous system disorders) | 0 | 4 | 0
Aggression (Psychiatric disorders) | 1 | 6 | 2
Irritability (Psychiatric disorders) | 3 | 5 | 2
Abnormal behaviour (Psychiatric disorders) | 0 | 4 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT02224703/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/03/NCT02224703/SAP_001.pdf